CLINICAL TRIAL: NCT03455413
Title: Electrical Impedance Tomography (EIT) in Assessing the Quality of Perioperative Invasive Ventilation in PICU
Brief Title: Quality of Perioperative Invasive Ventilation in PICU
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Other Study IDs: EETTMK:36/2017
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Invasive Ventilation; Elective Surgery
Keywords: electrical impedance tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Swisstom BB2 EIT device — Swisstom BB2 EIT device and NeoSensor Belts will be used to assess lung aeration, ventilation distribution and strech during invasive ventilation in perioperative care.

SUMMARY:
This is purely observational study in which quality of invasive ventilation is observed with electrical impedance tomography (EIT) during perioperative intensive care. EIT parameters will be used to assess if protective ventilation strategies are successfully followed during routine care.

DETAILED DESCRIPTION:
20 neonates and infants undergoing elective surgery and requiring postoperative treatment and follow up in PICU or in pediatric anestesiology clinic, will be included in this prospective observational study. Swisstom BB2-monitor and NeoSensorBelts will be used to monitor their ventilatory care from arrival to the operation room (prior intubation) to postoperative intensive care (until 2 hours after extubation). EIT parameters assessing lung aeration and ventilation distribution will be used to assess the quality of invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from a parent of legal guardian
* Infant undergoing elective or semi-elective surgery
* Postoperative admission to PICU expected
* Spontaneous breathing prior to study inclusion

Exclusion Criteria:

* Need for respiratory support prior to surgery
* Thoracic surgery
* Body weight < 1500g or > 10 kg

Ages: 2 Hours to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates and infants undergoing elective/semi-elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Silent spacies | 24 hours
  Amount of silent spaces observed in different phases of treatment in comparison to baseline

SECONDARY OUTCOMES:
Ventilation distribution | 24 hours
  Changes from baseline in ventilation distribution will be assessed in different phases of treatment
Effect of interventions on ventilatory parameters | 24 hours
  Relationship between intubation/invasive ventilation/extubation/spontaneous breathing and EIT findings

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kallio, MD, PhD, Study Director — Oulu University Hospital and PEDEGO research group, University of Oulu; Marika Rahtu, Principal Investigator — Oulu University Hospital and PEDEGO research group, University of Oulu
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No